CLINICAL TRIAL: NCT00172276
Title: Angiotensin Converting Enzyme Gene Polymorphism in Children With Idiopathic Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701241
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Aims This study was conducted to examine the association between the ACE insertion/deletion (I/D) genotype distribution in children with idiopathic nephrotic syndrome and the response to steroid therapy.

Patients and Methods The patients with idiopathic nephrotic syndrome were divided into 2 groups according to their clinical response to steroid: SS group including infrequent and frequent relapsers and non-SS group including steroid resistant (SR) and steroid dependent (SD) patients. Children without previous renal diseases and negative proteinuria were enrolled as control group in genetic study. The genotypes for ACE gene I/D polymorphism including DD, ID and II were analyzed by the newly developed automatic denaturing high performance liquid chromatography system (DHPLC).

ELIGIBILITY:
Inclusion Criteria:

* Total 59 children diagnosed as nephrotic syndrome at the age of 1 to 10 year-old were recruited in this study. These children with nephrotic syndrome were under follow-up at the Pediatric Nephrology Clinic in National Taiwan University Hospital. In addition, children without previous renal diseases and negative proteinuria were enrolled as control group in genetic study.

Ages: 1 Year to 10 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Kwei Tsau, MD, Principal Investigator — National Taiwan University Hospital